CLINICAL TRIAL: NCT05090020
Title: Systematic Review of Hypernatremia Following Hydatid Cyst Treatment
Brief Title: Hypernatremia in Hydatid Cyst Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trabzon Kanuni Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Aydın Aktaş, Associate Professor Doctor, Trabzon Kanuni Education and Research Hospital
Other Study IDs: TrabzonKERH
Record Dates: First submitted 2021-09-26; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Echinococcosis, Hepatic
Keywords: Echinococcosis; Hepatic; hypernatremia
MeSH Terms: conditions — Echinococcosis, Hepatic; Echinococcosis; Hypernatremia | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypernatremia: Hypernatremia (plasma sodium value above 145 mmol/L) due to HS use in the treatment of hydatid cyst.
  Interventions: Procedure: Treatment

INTERVENTIONS:
Procedure: Treatment — Surgery and PAIR

SUMMARY:
Hypertonic saline (HS) is one of the most widely used scolocidal agents in the treatment of hydatid cysts. Hypernatremia is one of the complications associated with the use of HS. It can cause hypernatremia, acid-base disorder, impaired lung, renal, cardiac and neurological functions and even death. Therefore, caution should be exercised in the use of HS, and open technique should be preferred in surgery.

ELIGIBILITY:
Inclusion Criteria: Patients who developed hypernatremia (plasma sodium value above 145 mmol/L) due to HS use in the treatment of hydatid cyst were included to study -

Exclusion Criteria:Patients who developed hypernatremia due to other treatments were excluded from the study.

-

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated who hydatid cyst with hypertonic saline
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Prevention of hypernatreima | 3 month
  Hypernatremia is plasma sodium value above 145 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Aydin Aktas, Study Chair — Kanuni Training and Research Hospital
Locations (1):
- Aydıin Aktas, Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No